CLINICAL TRIAL: NCT00022867
Title: Optimization of Calcium Absorption and Bone Formation During Early Puberty
Brief Title: Encouraging Calcium Absorption and Bone Formation During Early Puberty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AR043740 (NIH); R01AR043740 (NIH)
Record Dates: First submitted 2001-08-14; First posted 2001-08-16 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Bone growth; Calcium; Children; Diet; Puberty
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nondigestible oligosaccharide (NDO)

SUMMARY:
Increasing bone mass during puberty can ultimately decrease the risk of developing osteoporosis, which causes bones to weaken and break more easily later in life. The purpose of this study is to compare calcium absorption and bone growth in boys and girls on diets including either a nondigestible oligosaccharide (NDO) or simple sugar.

DETAILED DESCRIPTION:
Rapid increases in bone mass occur during calcium absorption and bone calcium deposition during puberty, and these increases can enhance peak bone mass and ultimately decrease the lifetime risk of osteoporosis. However, dietary, hormonal, and genetic factors likely affect increased bone mass. This study will examine if adding NDO to a pubertal diet allows more absorption of calcium by the body, producing stronger bones. The study will also assess how the hormones produced by the body during puberty affect bone growth and whether genetic factors affect calcium absorption or bone growth.

This study will last 2 years. At study entry, baseline pubertal hormone levels and bone mass will be assessed. Both a dual-energy X-ray absorptiometry (DEXA) scan and a calcium stable kinetic study measuring calcium absorption will be performed. Participants will then be randomly assigned to receive calcium fortified food with or without added NDO for 1 year. Calcium absorption will be measured again at 2 months. After the first year, calcium kinetic, hormonal, and DEXA studies will be performed and compared to baseline results. A final DEXA scan will be performed at the end of 2 years.

ELIGIBILITY:
* Tanner Stage 2 or 3
* Girls must not have started menstruating
* In the 10th to 90th percentile in body mass index (BMI) for their age

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center at Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Abrams SA, O'Brien KO. Calcium and bone mineral metabolism in children with chronic illnesses. Annu Rev Nutr. 2004;24:13-32. doi: 10.1146/annurev.nutr.24.012003.132135. PMID 15189111
- [Result] Abrams SA, Griffin IJ, Hawthorne KM, Liang L, Gunn SK, Darlington G, Ellis KJ. A combination of prebiotic short- and long-chain inulin-type fructans enhances calcium absorption and bone mineralization in young adolescents. Am J Clin Nutr. 2005 Aug;82(2):471-6. doi: 10.1093/ajcn.82.2.471. PMID 16087995
- [Result] Abrams SA, Griffin IJ, Hawthorne KM, Gunn SK, Gundberg CM, Carpenter TO. Relationships among vitamin D levels, parathyroid hormone, and calcium absorption in young adolescents. J Clin Endocrinol Metab. 2005 Oct;90(10):5576-81. doi: 10.1210/jc.2005-1021. Epub 2005 Aug 2. PMID 16076940
- [Result] Abrams SA, Griffin IJ, Hawthorne KM, Chen Z, Gunn SK, Wilde M, Darlington G, Shypailo RJ, Ellis KJ. Vitamin D receptor Fok1 polymorphisms affect calcium absorption, kinetics, and bone mineralization rates during puberty. J Bone Miner Res. 2005 Jun;20(6):945-53. doi: 10.1359/JBMR.050114. Epub 2005 Jan 31. PMID 15883634